CLINICAL TRIAL: NCT01621256
Title: Double-blind, Randomized, Placebo-controlled Study on Efficacy, Safety and Tolerability of Ancrod in Patients With Sudden Sensorineural Hearing Loss (SSHL)
Brief Title: Efficacy, Safety, and Tolerability of Ancrod in Patients With Sudden Hearing Loss
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nordmark Arzneimittel GmbH & Co. KG (Industry)
Collaborators: ClinSupport GmbH (Industry); MWI Medizinisches Wirtschaftsinstitut GmbH (Unknown); ProjectPharm s.r.o. (Unknown); LCR Leading Clinical Research s.r.o. (Unknown); X-act Cologne Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NM-V-101; 2012-000066-37 (EudraCT Number)
Record Dates: First submitted 2012-06-12; First posted 2012-06-18 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Hearing Loss; Deafness; Hearing Loss, Sensorineural; Hearing Disorders; Ear Diseases
MeSH Terms: conditions — Hearing Loss; Deafness; Hearing Loss, Sensorineural; Hearing Disorders; Ear Diseases | interventions — Ancrod; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ancrod (Experimental): Ancrod
  Interventions: Drug: Ancrod
- Saline solution (Placebo Comparator): Saline solution
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Ancrod — Day 1: Intravenous infusion; Days 2, 4, and 6: Subcutaneous injections
  Other Names: Viprinex; NM-V
  Arms: Ancrod
Drug: Saline solution — Day 1: Intravenous infusion; Days 2, 4, and 6: Subcutaneous injections
  Other Names: Placebo
  Arms: Saline solution

SUMMARY:
The purpose of this study is to determine whether ancrod is effective and safe in the treatment of sudden sensorineural hearing loss (SSHL).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral idiopathic sudden sensorineural hearing loss ≥30 dB
* Symmetric hearing prior to onset of SSHL
* Enrollment has to be accomplished within 7 days after SSHL onset

Exclusion Criteria:

* Bilateral SSHL
* Incomplete recovery after previous SSHL
* Previously existing, known retrocochlear hearing loss
* Any history of any ear operation or local inflammatory disease in the past one year
* History of blunt or penetrating ear trauma, head trauma, barotrauma, or acoustic trauma immediately preceding SSHL
* History of Meniere's disease, autoimmune hearing loss, radiation-induced hearing loss, endolymphatic hydrops.
* Treatment with steroids for any reason within the preceding 30 days.
* Body weight > 140 kg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-05; Primary Completion 2018-09-18 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Change in PTA (pure tone audiogram) in the affected ear | From baseline to Day 8

SECONDARY OUTCOMES:
Change in speech recognition in the affected ear | From baseline to Day 8

OTHER OUTCOMES:
Patient assessment of change in hearing impairment | From baseline to Day 8, Day 30 and Day 90
Change in fibrinogen concentration | From baseline to Day 2 and Day 8
Change in biomarkers | From baseline to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Martin Canis, MD PhD, Principal Investigator — Department for Otorhinolaryngology, LM University Munich
Locations (7):
- Czechia (2):
  - Site CZ, Hradec Králové
  - Site CZ, Prague
- Germany (5):
  - Site D, Göttingen
  - Site D, Hamburg
  - Site D, Hanover
  - Site D, Landsberg am Lech
  - Site D, München

IPD SHARING:
Plan to Share IPD: No